CLINICAL TRIAL: NCT01492504
Title: A Long-Term Follow-up Study of Subjects Who Participated in a Clinical Trial in Which Asunaprevir (BMS-650032) and/or Daclatasvir (BMS-790052) Was Administered for the Treatment of Chronic Hepatitis C
Brief Title: Three-year Follow-up Study of Subjects Who Participated in a Previous Asunaprevir (BMS-650032) and/or Daclatasvir (BMS-790052) Chronic Hepatitis C Clinical Trial
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: AI444-046; 2011-005287-21 (EudraCT Number)
Record Dates: First submitted 2011-11-30; First posted 2011-12-15 (Estimated); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — asunaprevir; daclatasvir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subjects with chronic hepatitis C: Subjects who participated in a clinical trial in which Asunaprevir (BMS-650032) and/or Daclatasvir (BMS-790052) was administered for the treatment of chronic hepatitis C
  Interventions: Drug: Asunaprevir (BMS-650032) and/or Daclatasvir (BMS-790052)

INTERVENTIONS:
Drug: Asunaprevir (BMS-650032) and/or Daclatasvir (BMS-790052) — Observational study - No Intervention [(subjects were previously treated with Asunaprevir (BMS-650032) and/or Daclatasvir (BMS-790052)]

SUMMARY:
The primary purpose of this study is to determine whether the hepatitis C virus continues to remain unable to be detected in subjects who were previously treated with Asunaprevir (BMS-650032) and/or Daclatasvir (BMS-790052) and achieved sustained virologic response.

ELIGIBILITY:
Inclusion Criteria

* Signed Written Informed Consent
* Subjects must have received at least one dose of Asunaprevir and/or Daclatasvir
* Subjects participating in Daclatasvir and/or Asunaprevir studies (ie, protocol numbers beginning with AI443, AI444 or AI447) may enroll regardless of virologic response
* Completed the required post-treatment follow-up period in previous study
* Must enroll in this study within 6 months of completing previous BMS study or within 6 months of protocol availability at the clinical site
* Men and women, ages 18 and older

Exclusion Criteria:

* Subject must not have been treated with any antiviral or immunomodulatory drug for chronic hepatitis C (CHC) after completion of the previous study during which Asunaprevir and/or Daclatasvir were administered
* Subject must not be participating in any other trial, excluding non-interventional trials
* Prisoners or subjects who are involuntarily incarcerated
* Subjects who are compulsorily detained for treatment of either a psychiatric or physical (eg, infectious disease) illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who participated in a clinical trial in which Asunaprevir (BMS-650032) and/or Daclatasvir (BMS-790052) was administered for the treatment of chronic hepatitis C
Sampling Method: Non-Probability Sample
Enrollment: 1850 (Estimated)
Dates: Start 2012-02-07 (Actual); Primary Completion 2018-03-16 (Actual); Study Completion 2018-03-19 (Actual)

PRIMARY OUTCOMES:
Durability of Sustained viral response [SVR] (time to loss of virologic response) | 24 or 48-week Intervals
  The durability of virologic response, as assessed by the time to loss of virologic response after achieving sustained viral response (SVR12) in a previous study with Asunaprevir (BMS-650032) and/or Daclatasvir (BMS-790052). Loss of virologic response assessed using Hepatitis C virus (HCV) Ribonucleic acid (RNA)

SECONDARY OUTCOMES:
Frequency of viral genotypic substitutions in subjects previously treated with Asunaprevir (BMS-650032) and/or Daclatasvir (BMS-790052) who did not achieve or did not maintain SVR12 | 24 or 48-week intervals
Long-term progression of liver disease, as measured by the frequency of hepatic disease progression, all cause mortality, and liver-related mortality | 24 or 48-week intervals

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (151):
- United States (50):
  - Alabama Liver & Digestive Specialists (Alds), Montgomery, Alabama
  - Pacific Oaks Medical Group, Beverly Hills, California
  - Southern California Research Center, Coronado, California
  - Scripps Clinic, La Jolla, California
  - Keck Medical Center of USC, HCC 1, Los Angeles, California
  - Peter J Ruane Md Inc, Los Angeles, California
  - Anthony M. Mills Md Inc, Los Angeles, California
  - Precision Research Institute, Llc, San Diego, California
  - Quest Clinical Research, San Diego, California
  - Medical Associates Research Group, San Diego, California
  - U.Cal.-San Francisco, San Francisco, California
  - University Of Colorado Denver & Hospital, Aurora, Colorado
  - Yale New Haven Hospital, New Haven, Connecticut
  - Schiff Center for Liver Diseases, Miami, Florida
  - University Of Miami School Of Medicine, Miami, Florida
  - Orlando Immunology Center, Orlando, Florida
  - Florida Hospital Transplant Center, Orlando, Florida
  - Gastrointestinal Specialists Of Georgia, Marietta, Georgia
  - Ruth M. Rothstein CORE Center, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - Mercy Medical Center, Baltimore, Maryland
  - Digestive Disease Associates, P.A., Catonsville, Maryland
  - Johns Hopkins University, Lutherville, Maryland
  - The Research Institute, Springfield, Massachusetts
  - University Of Michigan, Ann Arbor, Michigan
  - Saint Louis University, St Louis, Missouri
  - Southwest Care Center, Santa Fe, New Mexico
  - Nyu Medical Center, Great Neck, New York
  - University Of North Carolina At Chapel Hill School Of Med, Chapel Hill, North Carolina
  - Carolinas Medical Center, Charlotte, North Carolina
  - Carolinas Center For Liver Disease, Statesville, North Carolina
  - Mayo Clinic Rochester, Tulsa, Oklahoma
  - Healthcare Research Consultants, Tulsa, Oklahoma
  - Oregon Health & Science University, Portland, Oregon
  - Lehigh Valley Health Network, Allentown, Pennsylvania
  - University Of Pennsylvania School Of Medicine, Philadelphia, Pennsylvania
  - Gastro One, Germantown, Tennessee
  - Nashville Medical Research Institute, Nashville, Tennessee
  - Texas Clinical Research Institute, Arlington, Texas
  - Baylor College Of Medicine, Houston, Texas
  - Liver Associates Of Texas, Houston, Texas
  - MEDVAMC, Houston, Texas
  - Alamo Medical Research, San Antonio, Texas
  - Lifetree Clinical Research, Salt Lake City, Utah
  - Metropolitan Research, Annandale, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Bon Secours St. Mary's Hospital of Richmond, Inc., Richmond, Virginia
  - Mcguire Dvamc, Richmond, Virginia
  - Harborview Medical Center, Seattle, Washington
  - Ssm Health Dean Med Group, Madison, Wisconsin
- Argentina (6):
  - Fundacion Cidea De Paraguay, Ciudad de Buenos Aires, Buenos Aires
  - Centro Oncologico Integral, Mar del Plata, Buenos Aires
  - Hospital Austral, Prov. Buenos Aires, Buenos Aires
  - Instituto Centralizado De Asistencia E Investigacion Clinica, Prov de Santa Fe, Santa Fe Province
  - Local Institution, Buenos Aires
  - Hospital Italiano De Buenos Aires, Buenos Aires
- Australia (9):
  - Local Institution, Camperdown, New South Wales
  - Local Institution, Darlinghurst, New South Wales
  - Local Institution, Darlinghurst Nsw, New South Wales
  - Local Institution, Randwick, New South Wales
  - Local Institution, Westmead, New South Wales
  - Local Institution, Woollongabba, Queensland
  - Local Institution, Adelaide, South Australia
  - Local Institution, Clayton Vic, Victoria
  - Local Institution, Melbourne, Victoria
- Brazil (3):
  - Local Institution, Porto Alegre, Rio Grande do Sul
  - Local Institution, Rio de Janeiro
  - Local Institution, São Paulo
- Canada (7):
  - Local Institution, Calgary, Alberta
  - Local Institution, Edmonton, Alberta
  - Local Institution, Vancouver, British Columbia
  - Local Institution, Victoria, British Columbia
  - Local Institution, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Local Institution, Regina, Saskatchewan
- Denmark (2):
  - Local Institution, Hvidovre
  - Local Institution, Odense
- France (13):
  - Local Institution, Clichy
  - Local Institution, Créteil
  - Local Institution, La Roche-sur-Yon
  - Local Institution, Lille
  - Local Institution, Limoges
  - Local Institution, Lyon
  - Local Institution, Marseille
  - Local Institution, Montpellier
  - Local Institution, Nice
  - Local Institution, Paris
  - Local Institution, Pessac
  - Local Institution, Toulouse
  - Local Institution, Vandœuvre-lès-Nancy
- Germany (7):
  - Local Institution, Düsseldorf
  - Local Institution, Essen
  - Local Institution, Frankfurt
  - Local Institution, Hamburg
  - Local Institution, Hanover
  - Local Institution, Heidelberg
  - Local Institution, Mainz
- Ireland (2):
  - Mater Misericordiae University Hospital, Dublin, Dublin
  - St. James'S Hospital, Dublin, Dublin
- Italy (6):
  - Local Institution, Brescia
  - Local Institution, Cisanello (pisa)
  - Local Institution, Milan
  - Local Institution, Pavia
  - Local Institution, Torino
  - Local Institution, Viale Del Policlinico, 155
- Japan (24):
  - Local Institution, Nagoya, Aichi-ken
  - Local Institution, Chiba, Chiba
  - Local Institution, Fukuoka, Fukuoka
  - Local Institution, Kurume, Fukuoka
  - Local Institution, Ogaki-shi, Gifu
  - Local Institution, Hiroshima, Hiroshima
  - Local Institution, Sapporo, Hokkaido
  - Local Institution, Amagasaki-shi, Hyōgo
  - Local Institution, Kanazawa, Ishikawa-ken
  - Local Institution, Takamatsu, Kagawa-ken
  - Local Institution, Kagoshima, Kagoshima-ken
  - Local Institution, Kawasaki-shi, Kanagawa
  - Local Institution, Sendai, Miyagi
  - Local Institution, Okayama, Okayama-ken
  - Local Institution, Osaka, Osaka
  - Local Institution, Osaka-sayama-shi, Osaka
  - Local Institution, Suita, Osaka
  - Local Institution, Suita-shi, Osaka
  - Local Institution, Iruma-gun, Saitama
  - Local Institution, Bunkyo-ku, Tokyo
  - Local Institution, Minato-ku, Tokyo
  - Local Institution, Musashino-shi, Tokyo
  - Local Institution, Shinagawa-ku, Tokyo
  - Local Institution, Chuo-shi, Yamanashi
- Mexico (3):
  - Local Institution, Guadalajara, Jalisco
  - Local Institution, Cuernavaca, Morelos
  - Local Institution, Monterrey, Nuevo León
- Local Institution, Bialystok, Poland
- Local Institution, San Juan, Puerto Rico
- South Korea (2):
  - Local Institution, Yangsan, Gyeongsangnam-do
  - Local Institution, Busan
- Spain (7):
  - Local Institution, Alicante
  - Local Institution, Barcelona
  - Local Institution, Madrid
  - Local Institution, Málaga
  - Local Institution, Santiago de Compostela
  - Local Institution, Seville
  - Local Institution, Valencia
- Sweden (2):
  - Local Institution, Gothenburg
  - Local Institution, Stockholm
- Local Institution, Taichung, Taiwan
- United Kingdom (5):
  - Kings College Hospital, London, Greater London
  - Local Institution, London, Greater London
  - Imperial College London, London, Greater London
  - North Manchester General Hospital, Manchester, Greater Manchester
  - Gartnaval General Hospital, Glasgow

REFERENCES:
- [Derived] Reddy KR, Pol S, Thuluvath PJ, Kumada H, Toyota J, Chayama K, Levin J, Lawitz EJ, Gadano A, Ghesquiere W, Gerken G, Brunetto MR, Peng CY, Silva M, Strasser SI, Heo J, McPhee F, Liu Z, Yang R, Linaberry M, Noviello S. Long-term follow-up of clinical trial patients treated for chronic HCV infection with daclatasvir-based regimens. Liver Int. 2018 May;38(5):821-833. doi: 10.1111/liv.13596. Epub 2017 Oct 12. PMID 28941023
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/Pages/Investigator_inquiry_form.aspx